CLINICAL TRIAL: NCT05014048
Title: Vitamin D Supplementation for the Prevention of Acute Respiratory Tract Infection: a Randomized, Double-blinded and Plasebo Controlled Trial Among Young Finnish Men
Brief Title: Vitamin D Supplementation for the Prevention of Acute Respiratory Infections: a RCT in Young Finnish Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Finnish Defense Forces (Other Government)
Responsible Party: Principal Investigator, Ilkka Laaksi, Principal Investigator, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UTampere
Record Dates: First submitted 2020-12-16; First posted 2021-08-20 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Vitamin D Deficiency; Respiratory Tract Infections
MeSH Terms: conditions — Vitamin D Deficiency; Respiratory Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D3 (Active Comparator): 20 mikrog vitamin D3 daily, 3 months
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 20 mikrog vitamin D3 daily
  Arms: vitamin D3
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Vitamin D intervention effects on the prevention of acute respiratory tract infections among Young Finnish Men

ELIGIBILITY:
Inclusion Criteria;

* Male
* 18-29 years of age
* examined as Healthy according to Finnish Military Health Care regulations

Exclusion Criteria

* Female
* age > 30 yrs

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Days off duty due to acute respiratory tract infections | 4 months
  The number of Days off Duty recommended by Health care personnel will be calculated in order to show the severity and last of the disease. By that it could be estimated how the disease will effect on duty service.

SECONDARY OUTCOMES:
Days off duty due to musculoskeletal disorders | 4 months
  The number of days off Duty because of musculoskeletal disorders will be index for outcome. The index will be compared between plasebo and intervention group
Aerobic and muscular fitness | 4 months
  Used test are Cooper-test for aerobic and Finnish military fitness test for muscular fitness performance. The index will be compared between plasebo and intervention group

CONTACTS AND LOCATIONS:
Overall Officials: ilkka laaksi, MDPhD, Principal Investigator — University of Tampere, Finland
Locations (1):
- Finnish Defence Forces, Hämeenlinna, Finland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Laaksi A, Kyrolainen H, Pihlajamaki H, Vaara JP, Luukkaala T, Laaksi I. Effects of Vitamin D Supplementation and Baseline Vitamin D Status on Acute Respiratory Infections and Cathelicidin: A Randomized Controlled Trial. Open Forum Infect Dis. 2024 Aug 27;11(9):ofae482. doi: 10.1093/ofid/ofae482. eCollection 2024 Sep. PMID 39301110